CLINICAL TRIAL: NCT03265730
Title: Incidence, Risk Factors and Severity of Pediatric Antibiotic Associated Diarrhea
Brief Title: Pediatric Antibiotic Associated Diarrhea
Acronym: TURPENADA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ates Kara, Prof Dr, Hacettepe University
Other Study IDs: Hacettepe01
Record Dates: First submitted 2017-03-24; First posted 2017-08-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Diarrhea
Keywords: Outpatient clinics; oral antibiotics; diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diarrhea is one of the side effects of antibiotics. Antibiotic associated diarrhea can be encountered between two hours to two months after starting of antibiotics. The purpose of the study is to determine incidence,risk factors and severity of pediatric antibiotic associated diarrhea in Turkey.

DETAILED DESCRIPTION:
Antibiotic associated diarrhea is a common adverse effect, occurring about 5-30% of patients either early during treatment or up to two months after the cessation of the treatment. The frequency differs according to the definition of diarrhea, the inciting antimicrobial agent and the host factors such geriatric age, immunosuppression, prolonged hospitalization. Almost all agents, especially the the ones acting on anaerobes may cause diarrhea. Clinical presentations range from mild diarrhea to fulminant pseudomembranous enterocolitis. In Turkey still data about antibiotic associated diarrhea is not enough. Incidence and the factors that effect severity are not known.

ELIGIBILITY:
Inclusion Criteria:

* The parents and the child who give consent
* The children who are treated for the acute infections in the outpatient clinics and whole treatment is completed in the outpatient clinics.
* Children who are born mature, for the children who are younger than 1 year of age.

Exclusion Criteria:

* The parents and child who do not give consent
* Children who have primary and secondary immunosuppressive states.
* Children who had abdominal/gastrointestinal tract surgery in the past.
* Children who had used probiotics/prebiotics in the last one month period.
* Children who had used antibiotics in the last one month period.
* Children who has accompanying gastrointestinal symptoms.
* Children who are using anti-acid treatment at the time of involvement.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who admit to outpatient clinics and are ordered oral antibiotics for acute infections such as upper and lower respiratory tract infections, infections of mouth, urinary tract infections, skin and soft tissue infections.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Antibiotic Associated Diarrhea (AAD) in Children in Turkey | December 2018
  How common the antibiotic associated diarrhea is encountered in pediatric age group in outpatient clinic in Turkey.

SECONDARY OUTCOMES:
Local differences in pediatric AAD across Turkey | December 2018
  Differences in incidence and severity of AAD in children in different cities in Turkey.
  The incidence of antibiotic associated diarrhea will be expressed as proportion of new cases of diarrhea to total number of patients in the follow-up period of patients who receive oral antibiotics. The overall ratio will be calculated at the end of whole study period.
Follow-up of Severity of AAD in Outpatient Clinics and by Phone Calls for Two Months Period in Pediatric Population in Turkey. | December 2018
  Duration of AAD and interventional requirements of pediatric patients who develop AAD.
  Development of diarrhea during study period will be determined by using Bristol Stool Charts. Stool charts will be provided to parents by the investigators. The parents will follow number and shape and consistency of stool , and decide according to the Bristol Stool Chart. Four times and more defecation and stool in type 5,6 and 7 according to Bristol Chart that will continue for a minimum of 2 days will be regarded as diarrhea. If the diarrhea necessitates hospitalization and/or intravenous hydration therapy, this will be regarded as severe diarrhea. If patient with diarrhea will treated by just observation and diarrhea will subside spontaneously, diarrhea will be regarded as mild.
Incidence of antibiotic associated diarrhea with different type and formulation of antibiotic | December 2018
  Incidence of antibiotic associated diarrhea with different class of antibiotics will be determined
Incidence of antibiotic associated diarrhea in different age groups | December 2018
  Differences in incidence and severity of AAD in children with different age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ates Kara, Professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wistrom J, Norrby SR, Myhre EB, Eriksson S, Granstrom G, Lagergren L, Englund G, Nord CE, Svenungsson B. Frequency of antibiotic-associated diarrhoea in 2462 antibiotic-treated hospitalized patients: a prospective study. J Antimicrob Chemother. 2001 Jan;47(1):43-50. doi: 10.1093/jac/47.1.43. PMID 11152430
- [Background] Lau CS, Chamberlain RS. Probiotics are effective at preventing Clostridium difficile-associated diarrhea: a systematic review and meta-analysis. Int J Gen Med. 2016 Feb 22;9:27-37. doi: 10.2147/IJGM.S98280. eCollection 2016. PMID 26955289
- [Background] Barbut F, Meynard JL. Managing antibiotic associated diarrhoea. BMJ. 2002 Jun 8;324(7350):1345-6. doi: 10.1136/bmj.324.7350.1345. No abstract available. PMID 12052785
- [Background] Szajewska H, Canani RB, Guarino A, Hojsak I, Indrio F, Kolacek S, Orel R, Shamir R, Vandenplas Y, van Goudoever JB, Weizman Z; ESPGHAN Working Group for ProbioticsPrebiotics. Probiotics for the Prevention of Antibiotic-Associated Diarrhea in Children. J Pediatr Gastroenterol Nutr. 2016 Mar;62(3):495-506. doi: 10.1097/MPG.0000000000001081. PMID 26756877